CLINICAL TRIAL: NCT00035243
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Advanced Renal Cancer
Brief Title: EPO906 Therapy in Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2207; NCT00041002 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Neoplasms
Keywords: kidney cancer; renal cancer; cancer; tumor; tumour; neoplasm; carcinoma; clear cell; sarcomatoid; papillary; medullary; collecting duct; chromophobe; intravenous; epothilone
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms; Carcinoma | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: epothilone b

INTERVENTIONS:
Drug: epothilone b — EPO906 administered intravenously at 2.5 mg/m2 as a 5 minute bolus infusion repeated every week for three weeks followed by one week off The final tables and data is not in yet, so I cannot give you info on safety issues.

SUMMARY:
This study will examine whether the investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

The following patients may be eligible for this study:

* Histologically or cytologically documented evidence of epithelial renal cell carcinoma with at least one measurable lesion (if previous radiation treatment, the target lesion must have demonstrated progression since the radiation)
* Patients must have had a prior nephrectomy
* Must have a life expectancy of greater than three (3) months
* Patients who have had 0-1 prior cytokine treatment regimen (i.e. IL-2, IFN-?) or relapsed less than one year after such treatment may be eligible.

Exclusion Criteria:

The following patients are not eligible for this study:

* Patients who have received more than one (1) prior cytokine regimen (i.e. IL-2, IFN?) or relapsed more than one year after receiving such treatment are not eligible
* Patients who have had any prior chemotherapy (including a combination therapy)
* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports
* History of another malignancy within 3 years prior to study entry except curatively treated non-melanoma skin cancer, prostate cancer, or cervical cancer in situ
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* HIV+ patients
* Pregnant or lactating females.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-04; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST) | every 8 weeks

SECONDARY OUTCOMES:
Objective response rate (ORR) | every 8 weeks
Time to disease progression (TTP) | every 8 weeks
Overall Survival (OS) | every 8 weeks
Safety and tolerability of EPO906 | at each visit
Tumor-specific mutations and gene expression changes in tumor cells with blood cells and plasma | prior to the first treatment with EPO906, on the day of any clinically indicated tumor biopsy/resection and on the day of each tumor assessment
  For biomarker development

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - University of Maryland, Baltimore, Maryland
  - Wayne State University Karmanos Cancer Center, Detroit, Michigan
  - Our Lady Of Mercy Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Washington, Seattle, Washington
- France (2):
  - Centre L. Berard, Lyon
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=608